CLINICAL TRIAL: NCT02412891
Title: Evaluation of "UroShield" Device Impact Upon Side Effects and Complications of Urinary Catheter Usage
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancelled due to financial reasons
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0116-14-EMC
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Infectious
Keywords: introduction of urinary catheter
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients receive active UroShield device (Active Comparator): Patients receive active UroShield device
  Interventions: Device: UroShield device
- Patients receive inactive UroShield device (Sham Comparator): Patients receive inactive UroShield device
  Interventions: Device: Sham UroShield device

INTERVENTIONS:
Device: UroShield device — The UroShield device is Consists of two units:Actuator and Driver.
  Arms: Patients receive active UroShield device
Device: Sham UroShield device
  Arms: Patients receive inactive UroShield device

SUMMARY:
Evaluation of "UroShield" device impact upon side effects and complications of urinary catheter usage.

The use of urinary catheters is a common medical practice in the perioperative setting.

As such, it exposes the patient to certain comorbidities, including urinary tract infections.

The infectious process is known to begin with a development of a biofilm on the catheter's surface. This fact makes it an attractive target for UTI prevention technology.

Ultrasound waves were shown to reduce biofilm buildup in-vitro. We plan to determine the efficacy of this method in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need to insert a catheter urine as part of their treatment and rehabilitation at the orthopedic ward.

Exclusion Criteria:

1. Patients undergoing an invasive procedure in the past month some urinary tract, or the existence of a well-known structural pathology.
2. patients with a urinary tract infection in the past year.
3. Patients with a urinary tract infection when inserting a catheter.
4. pregnant women.
5. Patients under the age of 18.
6. without judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
side effects and complications of urinary catheter usage | One Year
  the measure is a composite of :complaints related to the uro-genital system, the results of blood and urine tests, monitoring fever, blood pressure and pulse